CLINICAL TRIAL: NCT00499460
Title: Modulation of Opioid Effects by Garlic Supplements
Brief Title: Effects of Garlic Supplements on Opioids in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Danny Shen, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2040.00; IR-6130 (Other: FHCRC IRB); CDR0000551927 (Other: PDQ); R21CA118334 (NIH)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Healthy, No Evidence of Disease
Keywords: Healthy, No Evidence of Disease
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Other): Two 30-day treatment periods separated by a washout of at least 4 weeks. In Period 1, participants receive oral garlic powder tablet twice daily on days 1-30, oral oxycodone on day 28, and a combination of oral midazolam and digoxin on day 29. In Period 2, participants receive oral placebo twice daily on days 1-30, oral oxycodone on day 28, and a combination of oral midazolam and digoxin on day 29.
  Interventions: Dietary Supplement: garlic powder tablets; Drug: oxycodone
- Arm II (Other): Two 30-day treatment periods separated by a washout of at least 4 weeks. In Period 1, participants receive oral placebo twice daily on days 1-30, oral oxycodone on day 28, and a combination of oral midazolam and digoxin on day 29. In Period 2, participants receive oral garlic powder tablet twice daily on days 1-30, oral oxycodone on day 28, and a combination of oral midazolam and digoxin on day 29.
  Interventions: Dietary Supplement: garlic powder tablets; Drug: oxycodone

INTERVENTIONS:
Dietary Supplement: garlic powder tablets — Each Garlicin tablet has a claimed allicin content of 3,200 microgram per tablet
  Other Names: Nature's Way Garlicin
Drug: oxycodone — Single administration of three 5-mg oxycodone tablets or a 15-mg dose
  Other Names: oxycodone hydrochoride, Roxicodone

SUMMARY:
RATIONALE: Garlic supplements may alter the pharmacokinetics of oxycodone, thereby affecting its effectiveness as an opioid analgesic for the relief of moderate or severe pain.

PURPOSE: This randomized phase 4 trial is studying how garlic supplements may change the pharmacokinetics of oxycodone and its analgesic and side effects in healthy volunteers.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether CYP3A (Cytochrome P450 3A) and/or P-glycoprotein mediated interactions exist between garlic supplements and oxycodone (a commonly used oral opioid analgesic) in healthy volunteers.

OUTLINE:

This is a single-blind, randomized, crossover study. Participants are randomized to 1 of 2 arms. Each arm entails two 30-day treatment periods, with a washout of at least 4 weeks in between.

* Arm I: In Period 1, participants receive oral garlic powder twice daily on days 1-28 and oral oxycodone on day 28. In Period 2, participants receive oral placebo twice daily on days 1-28 and oral oxycodone on day 28.
* Arm II: In Period 1, participants receive oral placebo twice daily on days 1-28 and oral oxycodone on days 28. In Period 2, participants receive oral garlic powder twice daily on days 1-28 and oral oxycodone on day 28.

In both periods of each arm, participants receive a combination of oral midazolam and oral digoxin for CYP3A and P-glycoprotein phenotyping on day 29. Blood samples are collected periodically and analyzed by liquid chromatography-mass spectrometry (LC-MS).

Blood and urine samples are collected after receiving oxycodone for pharmacokinetic characterization. Plasma concentrations of oxycodone and its metabolites are measured by LC-MS.

Response to experimentally induced pain by the Cold Pressor Test (CPT) is assessed at baseline and periodically after oxycodone treatment. Subjective ratings of opioid side effects are assessed by validated questionnaires for somatic side effects and cognitive function impairments.

ELIGIBILITY:
INCLUSION CRITERIA:

* Healthy volunteer
* Body mass index 20-32

EXCLUSION CRITERIA:

* Not pregnant
* No history of cardiopulmonary, liver, renal, endocrine, neurologic, or psychiatric disease
* No anemia
* No known adverse reactions to opioids, benzodiazepines, cardiac glycosides, or garlic supplements
* No known allergy or hypersensitivity to sulfur-containing food or drugs
* No significant gastrointestinal intolerance to lactose in dairy products
* No recent history of alcohol or substance abuse
* No history of or concurrent heavy daily consumption of allium vegetables (i.e., garlic, shallots, leeks, and chives)
* No handicaps due to visual and hearing impairments
* No resting heart rate < 50 beats per minutes
* No abnormal cardiac rhythm by EKG
* No unusually sensitive response or resistance to pain stimulation (Cold Pressor Test)
* Must be right handed
* No color blindness
* No history of learning disabilities or dyslexia
* Must be literate and proficient in English
* Must be a nonsmoker
* No concurrent medication except oral contraceptives
* No concurrent grapefruit or grapefruit juice
* No other concurrent over-the-counter herbal products or herbal tea

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2006-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danny D Shen, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was between November 2006 and August 2008. Healthy subjects were recruited from the University of Washington and Fred Hutchinson Cancer Research Center campuses through public notices.
Groups:
- Garlic First, Then Placebo: Two 30-day treatment periods separated by a washout of at least 4 weeks. In Period 1, participants receive oral garlic powder (Nature's Way Garlicin tablet) twice daily on days 1-30, and undergo testings with oxycodone on day 28 and a combination of oral midazolam and digoxin on day 29. In Period 2, participants receive oral placebo tablet twice daily on days 1-30, and undergo testings with oxycodone on day 28 and a combination of oral midazolam and digoxin on day 29.
- Placebo First, Then Garlic: Two 30-day treatment periods separated by a washout of at least 4 weeks. In Period 1, participants receive oral placebo tablet twice daily on days 1-30, and undergo testings with oxycodone on day 28 and a combination of oral midazolam and digoxin on day 29. In Period 2, participants receive oral garlic powder (Nature's Way Garlicin tablet) twice daily on days 1-30, and undergo testings with oxycodone on day 28 and a combination of oral midazolam and digoxin on day 29.
Period: Intervention 1 (30 Days)
Arm/Group | Garlic First, Then Placebo | Placebo First, Then Garlic
Started | 8 | 7
Completed | 6 | 7
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Fainting upon Blood Draw | 1 | 0
Period: Intervention 2 (30 Days)
Arm/Group | Garlic First, Then Placebo | Placebo First, Then Garlic
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Of the 15 enrollees, 6 subjects completed the study protocol in each assigned arm; hence, baseline analysis is only available in those 12 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Garlic First, Then Placebo | Placebo First, Then Garlic | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (5.2) | 30.5 (6.0) | 29.9 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Oxycodone Oral Clearance
Description: Oxycodone oral clearance is computed by Dose/AUC, where AUC is the area under the plasma oxycodone concentration-time curve from time zero to infinity. Oral clearance is a measure of the rate at which oxycodone is cleared from the body via metabolism.
Time Frame: Serial blood sampling over 24 hours after a 15-mg oral dose of oxycodone
Measure: Mean (Standard Deviation); unit: L/min
Groups:
- Garlic: Mean and standard deviation of oxycodone oral clearance following garlic powder treatment were calculated by pooling data from the active treatment period in each assigned arm
- Placebo: Mean and standard deviation of oxycodone oral clearance following placebo treatment were calculated by pooling data from the placebo treatment period in each assigned arm
Arm/Group | Garlic | Placebo
Number analyzed (Participants) | 12 | 12
L/min | 1.82 (0.40) | 2.04 (0.51)
Statistical Analysis 1: Comparison: Garlic vs Placebo; Test type: Superiority — The primary hypothesis being tested is that garlic powder treatment increases metabolic clearance of oxycodone through enzyme induction and results in lower exposure to oxycodone; p > 0.05, Generalized Estimating Equations — Significance probability for the treatment variable in the Generalized Linear Model; Response variable is oxycodone oral clearance. Explanatory variables include treatment, period and gender, along with their interaction terms

2. Secondary Outcome: Cold Pressor Tolerance AUC
Description: Cold Pressor Test measures response to experimentally induced pain, in this case by immersion of a subject's hand in icy-cold water. Tolerance is the duration of time a subject is able to keep his/her hand immersed in the cold water. A prolongation in tolerance time indicates analgesic response to oxycodone treatment. Cold Pressor Tolerance AUC is the area under the tolerance versus time curve over a 300-min period after a test dose of oxycodone. Because of non-normality in sample distribution, log transformed AUC estimates were analyzed by Generalized Linear Model.
Time Frame: Repeated testing for tolerance to Cold Pressor Test just before and at 45, 90, 150 and 300 min after a single 15-mg oral dose of oxycodone
Measure: Mean (Standard Deviation); unit: log (sec*min)
Groups:
- Garlic: Mean and standard deviation of Cold Pressor Test Tolerance AUC following garlic powder treatment were calculated by pooling data from the active treatment period in each assigned arm
- Placebo: Mean and standard deviation of Cold Pressor Test Tolerance AUC following placebo treatment were calculated by pooling data from the placebo treatment period in each assigned arm
Arm/Group | Garlic | Placebo
Number analyzed (Participants) | 12 | 12
log (sec*min) | 3.513 (0.904) | 3.715 (0.604)
Statistical Analysis 1: Comparison: Garlic vs Placebo; Test type: Superiority — The secondary hypothesis being tested is that powder garlic treatment lowers Cold Pressor Test tolerance (i.e., diminished analgesic response) after oxycodone administration due to a more rapid metabolic clearance and lower exposure to oxycodone; p > 0.05, Generalized Estimating Equations — Significance probability for the treatment variable in the Generalized Linear Model; Response variable is log Tolerance AUC. Explanatory variables include treatment, period and gender, along with their interaction terms

3. Secondary Outcome: Somatic Side Effects Total Score
Description: Subjects rated the bodily side effects they experienced at 90, 150 and 300 min after oxycodone administration on a 35-item Somatic Side Effects (SSE) questionnaire. Total score (i.e., average of the scores for all 35 items) ranges on a numerical scale from 0 (no somatic side effects) to a maximum of 4 (extreme somatic aide effects). Only the peak SSE scores at 150 min are reported herein.
Time Frame: SSE scores at 150 min after a single 15-mg oral dose of oxycodone
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Garlic: Mean and standard deviation of SSE Total Score following garlic powder treatment were calculated by pooling data from the active treatment period in each assigned arm
- Placebo: Mean and standard deviation of SSE Total Score following placebo treatment were calculated by pooling data from the placebo treatment period in each assigned arm
Arm/Group | Garlic | Placebo
Number analyzed (Participants) | 12 | 12
units on a scale | 0.560 (0.140) | 0.711 (0.184)
Statistical Analysis 1: Comparison: Garlic vs Placebo; Test type: Superiority — The secondary hypothesis being tested is that garlic powder treatment lowers opioid side effects after oxycodone administration due to a more rapid metabolic clearance and lower exposure to oxycodone; p > 0.05, Generalized Estimating Equations — Significance probability for the treatment variable in the Generalized Linear Model; Response variable is total SSE rating score. Explanatory variables include treatment, period, time and gender, along with their interaction terms

4. Secondary Outcome: Cognitive-Affective Side Effects Total Score
Description: Subjects rated the mental side effects they experienced at 90, 150 and 300 min after oxycodone administration on a 36-item Cognitive-Affective Side Effects (CASE) questionnaire. Total score (i.e., average of the scores for all 36 items) ranges on a numerical scale from 0 (no somatic side effects) to a maximum of 4 (extreme somatic aide effects). Only the peak CASE scores at 150 min are reported herein.
Time Frame: CASE scores at 150 min after a single 15-mg oral dose of oxycodone
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Garlic: Mean and standard deviation of CASE Total Score following garlic powder treatment were calculated by pooling data from the active treatment period in each assigned arm
- Placebo: Mean and standard deviation of CASE Total Score following placebo treatment were calculated by pooling data from the placebo treatment period in each assigned arm
Arm/Group | Garlic | Placebo
Number analyzed (Participants) | 12 | 12
units on a scale | 1.884 (0.118) | 1.714 (0.147)
Statistical Analysis 1: Comparison: Garlic vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p > 0.05, Generalized Estimating Equations — Significance probability for the treatment variable in the Generalized Linear Model; Response variable is total CASE rating score. Explanatory variables include treatment, period, time and gender, along with their interaction terms

5. Secondary Outcome: Oral Midazolam Test
Description: Midazolam when given orally is a probe substrate for the in vivo intestinal and hepatic activity of CYP3A (Cytochrome P450 3A) enzymes. The phenotype index in this case is the area under the plasma midazolam concentration from time zero to 360 min after a 5-mg oral test dose. A decrease in oral midazolam AUC indicates enhanced activity of CYP3A enzymes, possibly as a result of enzyme induction.
Time Frame: Serial blood sampling over 6 hours after a 5-mg oral test dose of midazolam
Measure: Mean (Standard Deviation); unit: (ng/mL)*min
Groups:
- Garlic: Mean and standard deviation of oral midazolam AUC following garlic powder treatment were calculated by pooling data from the active treatment period in each assigned arm
- Placebo: Mean and standard deviation of oral midazolam AUC following placebo treatment were calculated by pooling data from the placebo treatment period in each assigned arm
Arm/Group | Garlic | Placebo
Number analyzed (Participants) | 12 | 12
(ng/mL)*min | 2491 (789) | 2495 (825)
Statistical Analysis 1: Comparison: Garlic vs Placebo; The secondary hypothesis being tested is that garlic powder induces CYP3A-mediated metabolism resulting in a lower oral midazolam AUC; Test type: Superiority; p > 0.05, t-test, 1 sided; Garlic powder versus placebo

6. Secondary Outcome: Oral Digoxin Test
Description: Digoxin when given orally is a probe substrate for the efflux activity of P-glycoprotein in the small intestine. The phenotype index in this case is the area under the plasma digoxin concentration from time zero to 240 min after a 0.5-mg oral test dose. A decrease in oral digoxin AUC indicates an enhanced activity of P-glycoprotein, possibly as a result of transporter upregulation.
Time Frame: Serial blood sampling over 4 hours after a 0.5-mg oral test dose of digoxin
Measure: Mean (Standard Deviation); unit: (ng/mL)*min
Groups:
- Garlic: Mean and standard deviation of oral digoxin AUC following garlic powder treatment were calculated by pooling data from the active treatment period in each assigned arm
- Placebo: Mean and standard deviation of oral digoxin AUC following placebo treatment were calculated by pooling data from the placebo treatment period in each assigned arm
Arm/Group | Garlic | Placebo
Number analyzed (Participants) | 12 | 12
(ng/mL)*min | 231 (50) | 226 (58)
Statistical Analysis 1: Comparison: Garlic vs Placebo; Test type: Superiority — The secondary hypothesis being tested is that garlic powder treatment induces intestinal P-glycoprotein, reduces the bioavailability and hence AUC of orally administered digoxin; p > 0.05, t-test, 1 sided; Garlic powder versus placebo

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from all enrolled subjects over the 3-month duration of their study.
Description: Adverse event collection relied on subject self-reporting during the 30-day garlic or placebo treatment. Subjects were monitored by pulse oximetry and observed for opioid side effects by trained nurses on the oxycodone test day. Blood pressure and heart rate were monitored on the oral digoxin and midazolam test day.
Groups:
- Garlic: Data for all subjects during their active garlic treatment period in both arms were pooled.
- Placebo: Data for all subjects during their placebo treatment period in both arms were pooled.
Arm/Group | Garlic | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No